CLINICAL TRIAL: NCT04624529
Title: Validity and Reliability of a Self-evaluation Tool for Cognitive Deficits in the Acute Stage After Stroke
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Annick Van Gils, PhD, KU Leuven
Other Study IDs: S64120
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Stroke, Acute; Cognitive Dysfunction
Keywords: Occupational therapy; Evaluation tool
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self evaluation tool — This self-evaluation tool to evaluate cognitive function, developed by the occupational therapy department, is a paperwork task with guidelines for semi-structured interpretation.

SUMMARY:
Cognitive disorders are common early after stroke but can be overseen in patients with mild stroke who seem to be functionally recovered but are at risk to experience difficulties in advanced daily activities affecting social, vocational and family responsibilities. Acute stroke units admit a large number of patients and adequate referral to rehabilitation services is essential in terms of quality of care. A self-evaluation tool to evaluate cognitive function was developed by the occupational therapy department.

Patients with mild strokes and pre-stroke independent for instrumental daily activities fill out this self-evaluation tool, which is a paperwork task. Semi-structured interpretation is performed by physician and may result in referral to the occupational therapist for comprehensive evaluation.

In this study the validity and reliability of the self-evaluation tool will be examined.

ELIGIBILITY:
Inclusion Criteria:

* diagnose of stroke
* written consent
* age 18 years or older
* less than 1 week after stroke onset

Exclusion Criteria:

* not able to write/read
* not able to understand Dutch
* unilateral motor deficit in upper limb (NIHSS score for upper limb +2)
* referred to stroke unit with Transcient Ischemic Attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with stroke admitted to the acute stroke unit are consecutive recruited.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Self-evaluation tool | within one week after stroke onset
  cognitive screening tool
Oxford Cognitive Screen | within one week after stroke onset
  cognitive measure
Montreal Cognitive Assessement | within one week after stroke onset
  cognitive measure

CONTACTS AND LOCATIONS:
Overall Officials: Robin Lemmens, PhD, MD, Principal Investigator — UZ/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No